CLINICAL TRIAL: NCT01352065
Title: Phase 3 Characterization and Detection of Prolonged Endothelin Receptors Antagonists Administration
Brief Title: Characterization and Detection of Prolonged Endothelin Receptors Antagonists Administration
Acronym: ERAATH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Center for Health Sciences, Serbia (Other)
Responsible Party: Center for Health, Exercise and Sport Sciences, Serbia, Center for Health, Exercise and Sport Sciences, Serbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CHS-ERA-2011
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Pulmonary Hypertension
Keywords: Pharmacokinetics; Exercise performance; Athletes
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Bosentan; ambrisentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BOSENTAN (Experimental)
  Interventions: Drug: Bosentan
- AMBRISENTAN (Experimental)
  Interventions: Drug: Ambrisentan
- PLACEBO (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bosentan — tablet, 250 mg per day, twice per day, 8 weeks
  Arms: BOSENTAN
Drug: Ambrisentan — tablet, 10 mg per day, single per day, 8 weeks
  Arms: AMBRISENTAN
Drug: Placebo — Tablet, 10 mg per day, single per day, 8 weeks
  Arms: PLACEBO

SUMMARY:
Endothelin receptors antagonists (ERA), such as bosentan and ambrisentan, are a class of vasoactive drugs that have been developed for the treatment of pulmonary arterial hypertension. It has been anecdotally reported that ERA is frequently used among top-level athletes to counteract exercise-induced rise in pulmonary vascular pressures and increase exercise performance. Yet, the effects of ERA on exercise capacity in healthy humans are puzzling, with the drugs not included in the current Prohibited List, since the ergogenic potential is yet to be fully understood and determined. Furthermore, the urinary excretion of ERA metabolites following administration has not been studied systematically at rest and during exercise in athletes, as a way to detect its intake if performance-enhancing potential is confirmed. In the planned study ERA will be administered in newly approved doses for 8 weeks in order to assess the presumed doping potential for both male and female athletes, and to monitor serum and urinary ERA excretion dynamics after single- and multiple-dose administration. The possible effects of prolonged ERA administration in higher doses on exercise performance may be relevant, if further confirmed, in terms of their possible fraudulent utilization to influence exercise performance in sports, raising the difficult question of whether, particularly in some circumstances, the ERA might be considered as prohibited substances in athletes.

DETAILED DESCRIPTION:
Preliminary findings of our research group indicated that ERA enhances exercise performance (particularly aerobic) after 7-day intake of higher doses of non-selective ERA bosentan (doses used were approved for pulmonary arterial hypertension treatment). This is in part in accordance with results of previous research (Faoro et al. 2009), although authors administered regular single dose (62.5 mg) of bosentan in hypoxic healthy subjects. Our study should examine metabolic profiles of athletes after receiving significantly higher doses of two oral ERA as compared to previous research, along with assessment of ergogenic potential with 8 weeks of administration in placebo-control and randomized design. We expect that ERA will increase time to exhaustion during endurance test, increase the maximal oxygen uptake and rate of ultra-short term heart rate recovery after exercise, and affecting blood and urine cortisol, testosterone and dehydroepiandrosterone following administration. Moreover, we will clearly evaluate 24-h pharmacokinetic profile of ERA in blood and urine and collect data for concentration-time profiles of ERA and main active metabolites, in aim to provide more rationale basis for identification and detection for doping control.

ELIGIBILITY:
Inclusion Criteria:

* male and female volunteers
* experienced in athletic training (> 5 years of experience)
* aged 20 to 30 years
* free from musculoskeletal dysfunctions
* free from metabolic and heart diseases

Exclusion Criteria:

* pregnancy
* use of hormonal contraceptives
* use of dietary supplement that contains any ergogenic agent

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake | Change from Baseline in Maximal oxygen uptake at 8 weeks
  Maximal oxygen uptake is the maximum capacity of an individual's body to transport and use oxygen during incremental exercise, which reflects the physical fitness of the individual.

SECONDARY OUTCOMES:
Plasma concentration of bosentan | Regular sampling will be performed during administration at 0, 1, 2, 4, 6, and 8 weeks, and after 2 and 4 weeks post-administration

CONTACTS AND LOCATIONS:
Overall Officials: Sergej M Ostojic, MD, PhD, Study Director — Center for Health, Exercise and Sport Sciences
Locations (1):
- Center for Health, Exercise and Sport Sciences, Belgrade, Serbia

REFERENCES:
- [Derived] Ostojic SM, Stojanovic M, Calleja-Gonzalez J, Olcina G, Sekulic D, Hoffman JR. Performance-enhancing effects of non-selective endothelin receptor antagonist. Int J Cardiol. 2014 Feb 1;171(2):294-7. doi: 10.1016/j.ijcard.2013.11.077. Epub 2013 Dec 4. No abstract available. PMID 24342407